CLINICAL TRIAL: NCT05931276
Title: CSP #2026 - Beta Blocker Dialyzability on Cardiovascular Outcomes (BRAVO)
Brief Title: CSP #2026 - Beta Blocker Dialyzability on Cardiovascular Outcomes
Acronym: BRAVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026
Record Dates: First submitted 2022-03-29; First posted 2023-07-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: End-Stage Kidney Disease; End-Stage Renal Disease
Keywords: Dialysis; beta-Blockers, Adrenergic; Cardiovascular Diseases; Point of Care Research; Comparative Effectiveness Research; Metoprolol Succinate; Carvedilol; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Metoprolol; Carvedilol

STUDY DESIGN:
Intervention Model Description: The study design is a multicenter clinically integrated prospective randomized open-label blinded-endpoint (PROBE) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoprolol Succinate (Active Comparator): Depending on baseline type and dose of beta blocker:
  * 25 mg once daily (12.5 mg once daily if > NYHA class II)
  * 50 mg (or 25 mg) once daily
  * 100 mg (or 50 mg) once daily
  * 200 mg (or 100 mg titrated to 200 mg) once daily
  Interventions: Drug: Metoprolol Succinate
- Carvedilol (Active Comparator): Depending on baseline type and dose of beta blocker:
  * 3.125 mg twice daily
  * 6.25 mg twice daily
  * 12.5 mg twice daily
  * 25 mg twice daily (may titrate to 5 0mg twice daily if > 85 kg)
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Metoprolol Succinate — a dialyzable, beta-1 selective beta blocker
  Arms: Metoprolol Succinate
Drug: Carvedilol — a non-dialyzable, non-selective beta blocker with alpha-1 antagonist properties
  Arms: Carvedilol

SUMMARY:
The investigators aim to determine, using a point-of-care randomized controlled trial design, if hemodialysis patients, who are randomized to metoprolol succinate (a dialyzable, beta-1 selective beta blocker), have an improved cardiovascular outcome compared to those randomized to carvedilol (a non-dialyzable, non-selective beta blocker with alpha-1 antagonist properties). The investigators will also examine intervention practices to identify components that best support engagement and sustainability.

DETAILED DESCRIPTION:
Approximately 35,000 Veterans have end stage kidney disease (ESKD) with an incidence of 13,000 annually. These numbers are increasing because of the epidemic of diabetes, the most common cause of ESKD, among the Veteran population. Patients with ESKD on hemodialysis have substantial cardiovascular morbidity. Veterans annual mortality is in excess of 15% and more than half the deaths are due to cardiovascular disease. Beta blockers have been shown to prevent cardiovascular events in randomized clinical trials in patients without chronic kidney disease, particularly those with heart failure and after myocardial infarction. Beta blockers are a mainstay of therapy in dialysis patients, with two-thirds of Veterans on dialysis receiving a beta blocker. There are no head-to-head randomized studies comparing the two most commonly used beta blockers in ESKD patients in the United States, metoprolol and carvedilol, but observational studies suggest superior outcomes for patients treated with metoprolol. The identification of the superior beta blocker may significantly improve the morbidity and mortality of the VA dialysis population.

The investigators aim to compare two beta blockers with similar indications, usage and availability within the VA but with major differences in patients dialysis clearance and adrenergic effects. The investigators aim to determine if patients undergoing dialysis have improved survival when using metoprolol succinate, a beta blocker that is removed by dialysis and is beta-1 selective, compared to carvedilol, a beta blocker that is not removed by dialysis and is not beta-selective and is also an alpha-blocker.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis
* Received one of the following beta blockers through the VA pharmacy: metoprolol (succinate or tartrate), atenolol, labetalol, carvedilol, bisoprolol

Exclusion Criteria:

* Impaired decision-making capacity
* Patients not receiving carvedilol who have a history of asthma
* known hypersensitivity to any component of either drug
* Provider unwilling to sign a new medication order for a randomized patient
* No surrogate consent will be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2540 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to major cardiovascular event | Randomization to time to event; average follow-up 3 years
  The Primary outcome measure will be time to a non-fatal adverse cardiovascular event, defined as a composite outcome comprised of the first occurrence after randomization of any of the following: myocardial infarction, stroke, or hospitalization for heart failure, and all-cause mortality

SECONDARY OUTCOMES:
Non-fatal myocardial infarction | Randomization to time to event; average follow-up 3 years
  Non-fatal myocardial infarction
Non-fatal stroke | Randomization to time to event; average follow-up 3 years
  Non-fatal stroke
Hospitalization for heart failure | Randomization to time to event; average follow-up 3 years
  Hospitalization for heart failure
All-cause mortality | Randomization to time to event; average follow-up 3 years
  All-cause mortality

OTHER OUTCOMES:
All-cause hospitalization | Randomization to time to event; average follow-up 3 years
  All-cause hospitalization
ED visit or hospitalization possibly related to low BP including falls, fractures, hypotension, or serious injury | Number of events; average follow-up 3 years
  Number of emergency department visits or hospitalization for events that may be a consequence of low blood pressure or beta blocker excess or withdrawal including falls, fractures, hypotension, or serious injury
Use of BP raising medications | Use of drug; average follow-up 3 years
  Use and dose of midodrine
ED or hospital visits for atrial fibrillation and uncontrolled rate | Randomization to time to event; average follow-up 3 yars
  Emergency department visit or hospitalization for atrial fibrillation with uncontrolled rate (to capture poor control with beta blocker withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Areef Ishani, MD MS, Study Chair — Minneapolis VA Health Care System, Minneapolis, MN
Locations (8):
- United States (8):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leatherman SM, Ishani A. Point-of-Care Clinical Trials in Nephrology. J Am Soc Nephrol. 2024 Jun 1;35(6):812-814. doi: 10.1681/ASN.0000000000000340. Epub 2024 Feb 29. No abstract available. PMID 38419159